CLINICAL TRIAL: NCT05959733
Title: Maximal Repair Versus Bridging Reconstruction with BioBrace® for the Treatment of Chronic, Massive Rotator Cuff Tears: Clinical, Radiographic, and In-vivo Biomechanical Analysis
Brief Title: Maximal Repair Versus Bridging Reconstruction with BioBrace®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Principal Investigator, Ivan Wong, MD, MD Orthopaedic Surgeon, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BioBridge
Record Dates: First submitted 2023-07-05; First posted 2023-07-25 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Tears; Bioinductive Implant
Keywords: shoulder; rotator cuff; clinical outcomes; radiographic outcomes; biomechanics; bridging reconstruction; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware to the type of surgery that they received. The investigator will not be blinded, however, the individuals assessing the outcomes will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Repair (Active Comparator): This group will undergo a rotator cuff repair procedure.
  Interventions: Procedure: Repair
- Bridging Reconstruction using BioBrace (Experimental): This experimental group will undergo bridging reconstruction using the bioinductive implant, BioBrace.
  Interventions: Procedure: Bridging Reconstruction using BioBrace

INTERVENTIONS:
Procedure: Bridging Reconstruction using BioBrace — Patients in the reconstruction group will undergo maximal repair with interposition bridging using BioBrace. This technique will follow a previously described technique by the principal investigator with differences allocated to the graft, it's preparation and insertion. The bursa will be debrided, and rotator cuff edged will be shaved down to stable tissue. BioBrace is bioinductive scaffold composed of highly porous type I collagen and bio-resorbable poly (L-lactide) (PLLA) microfilaments, and will be used as the graft in this trial.
  Arms: Bridging Reconstruction using BioBrace
Procedure: Repair — Patients in the maximal repair group will undergo a SCOI-row rotator cuff repair with adequate tension as described previously, with recreation of the rotator cable. Briefly, the SCOI-row rotator cuff repair uses one triple loaded suture anchor for each 1.2cm of torn tendon. This technique has been completed in a previous randomized controlled trial.
  Arms: Repair

SUMMARY:
The purpose of this study is to determine if using BioBrace® to reconstruct the gap in the rotator cuff tears lead to better results for patients compared to the traditional maximal repair method. This study will use a variety of clinical, radiographic, and functional outcome measures. Specifically, the researchers will be comparing the re-tear rate, patient reported outcomes, shoulder strength, range of motion, muscle activation, in-vivo biomechanics, and other radiographic outcomes using x-ray and MRI.

ELIGIBILITY:
Inclusion Criteria:

* magnetic resonance imaging (MRI) proven diagnosis of a large or massive (> 3cm), two-tendon (supraspinatus and infraspinatus) tear of the shoulder rotator cuff
* over 18 years of age

Exclusion Criteria:

* glenohumeral osteoarthritis
* Western Ontario rotator cuff score >60
* uncontrolled diabetes (Hgb A1C >7%)
* pregnant
* local or systemic infection
* inability to cooperate with and/or comprehend post-operative instructions
* MRI proven non-vascular sites
* poor nutritional state (Alb <30 g/L)
* cancer
* paralysis of the shoulder
* contracture of the shoulder
* patients unable to provide informed consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic or clinical failure | 2 years
  The primary outcome measure for this study will be radiographic and/or clinical failure defined as a rotator cuff tear of equal or larger size than at baseline or does not meet WORC score MCID compared to baseline at any follow up

SECONDARY OUTCOMES:
Acromiohumeral Distance | 2 year
  Acromiohumeral distance (AHD) will be measured on pre- and post-operative x-rays.
Muscle Atrophy | 2 year
  Using MRI, muscle atrophy will be measured using Warner's classification between groups.
Fatty Infiltration | 2 year
  Fatty infiltration using the Goutallier classification will be used and identified
Healing Rate | 2 year
  To measure the structural integrity of the surgery, Sugaya method will be used.
Western Ontario Rotator Cuff Index (WORC) | Baseline, 6-month, 1-year, 2-years
  WORC will be measured pre-operatively, and post-operatively and 6-months, 1-year, and 2-years
American Shoulder and Elbow Surgeon survey | Baseline, 6-month, 1-year, 2-years
  American Shoulder and Elbow Surgeon survey will be measured pre-operatively, and post-operatively and 6-months, 1-year, and 2-years
EQ-5D-5L | Baseline, 6-month, 1-year, 2-years
  EQ-5D-5L for overall health will be measured pre-operatively, and post-operatively at 6-months, 1-year, and 2-years
Range of motion | Baseline, 6-month, 1-year, 2-years
  The range of motion, measured in degrees for flexion, extension, abduction, internal, and external rotation will be measured. These are measured and compared pre-operatively, and post-operatively and 6-months, 1-year, and 2-years
Shoulder strength | Baseline, 6-month, 1-year, 2-years
  The strength of patients flexion, extension, abduction, internal, and external rotation will be measured. These are measured and compared pre-operatively, and post-operatively and 6-months, 1-year, and 2-years
Biomechanics and Muscle Activity | Baseline and 2 years
  Pre- and post-operative (1-year) in-vivo biomechanics and electromyography will be compared between groups during a standardized shoulder lifting study in a laboratory based environment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wong, MD, Principal Investigator — Nova Scotia Health Authority, Orthopaedic Surgeon
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No